CLINICAL TRIAL: NCT04114396
Title: Investigating Poor Response to Monoclonal Therapy in Asthma
Brief Title: Poor Response to Monoclonal Therapy in Asthma
Acronym: PROCLAIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 18048
Record Dates: First submitted 2019-03-14; First posted 2019-10-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: Severe Asthma; Anti-IL5; Asthma
MeSH Terms: conditions — Asthma | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Viral throat swab
  2. Venous blood sampling: 40ml
  3. Bronchoscopy: 20 mls bronchial wash, 4 bronchial brushes, 6 bronchial biopsies
  4. Nasal brush
  5. Passive saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe asthma: Untreated by anti-IL5 treatment for severe asthma at point of recruitment. To be prescribed anti-IL5 as part of their treatment following consent. Note: Anti-IL5 treatment is prescribed as per agreed multidisciplinary team meeting, outside of the decision to enrol the patient on the study, and is administered by the clinical team as part of the patient's clinical care outside of the research study.
  Interventions: Drug: Anti-IL5 Antibody; Procedure: Bronchoscopy
- Healthy control: Control group without respiratory condition
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Drug: Anti-IL5 Antibody — Asthma group: Anti-IL5 treatment Control group: No biologic.
  Groups: Severe asthma
Procedure: Bronchoscopy — Optional for both arms

SUMMARY:
Asthma affects 8% of the entire population. 4-5% of asthma sufferers have severe asthma, characterised by recurrent exacerbations (worsening of symptoms leading to the person having a bout of corticosteroids and/or antibiotics), significant symptoms and lack of response to the most widely used therapy, corticosteroids.

There is now new types of treatments (antibody drugs) which are licensed to manage severe asthma such as Anti-IL5. There is evidence Anti-IL5 and other similar antibody drugs are effective at reducing asthma exacerbations and reduce the need for oral corticosteroids for those that have severe asthma.

However, some patients respond poorly to Anti-IL5 and the investigators would like to find out why this happens. It is hoped that the investigators can identify the mechanism of poor treatment response to Anti-IL5. It is also hoped that the investigators can understand why symptoms worsen to the point of requiring antibiotics and/or steroids (also known as an exacerbation) for those prescribed Anti-IL5.

ELIGIBILITY:
Inclusion criteria: case participants:

* Aged 18 - 80 years old
* Able to give informed consent
* All patients identified as being suitable for anti-IL5 therapy by the asthma MDT will be considered for study enrolment.

This assessment by the MDT for participants to be eligible includes:

* A measure of compliance with current asthma medication,
* Confirmation of asthma diagnosis
* Suitability for anti-IL5 therapy based on blood eosinophil counts,
* Asthma exacerbation rates
* Prednisolone dose.
* Confirmation of treatment requires at least two asthma specialists to agree that this is the correct course of action
* Patients must first demonstrate over 75% compliance with inhaled and/or oral corticosteroid therapy

The asthma MDT and difficult asthma clinic normally assess patients between 18-80 years so only patients in this age range will be approached.

All patients will be able to give informed consent for study participation.

Exclusion criteria: case participants:

• Pregnancy

Inclusion criteria: control participants:

* Aged between 18-80 years old.
* Able to give informed consent

Exclusion criteria: control participants:

* Pregnancy
* Underlying respiratory conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the severe asthma clinic. Once the multidisciplinary team (MDT) have decided that the patient will be prescribed anti-IL5 therapy a patient information sheet (PIS) will be posted out by the clinical team. If the appointment with the clinical team is within days of the MDT, potential participant will be approached by a member of the research team and the study will be discussed and a patient information sheet will be given to the patient.
  Control participants will be recruited from our Respiratory Research Database and have agreed to be contacted for research. A poster will be created to be put up in Nottingham City Hospital, Queen's Medical Centre and at the University of Nottingham, UK.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-12-31 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Identification of mechanisms associated with poor response to anti-IL5 therapy | 12 months
  Identification of mechanisms associated with poor response to anti-IL5 therapy. A poor response is defined as an inability to halve the pre-treatment annualised exacerbation rate; an asthma exacerbation is defined as a worsening of asthma symptoms necessitating a short burst of oral corticosteroids, or a doubling of maintenance oral corticosteroid treatment dose.
An improvement in FEV1 as assessed by spirometry | 12 months
  Treatment response as assessed as a clinically meaningful improvement in asthma control (ACQ change of >0.5).
A clinically meaningful improvement in asthma control as assessed by ACQ | 12 months
  An improvement in FEV1 of >100ml using spirometry.

SECONDARY OUTCOMES:
The identification of exacerbation pathogenesis in patients receiving anti-IL5 therapy via cytokine analysis | 12 months
  Blood cytokine analysis (analysed by Bio-plex 200 system) will be analysed at ad-hoc exacerbation visits to identify exacerbation pathogenesis.
The identification of exacerbation pathogenesis in patients receiving anti-IL5 therapy via viral throat swab analysis | 12 months
  Viral throat swabs results (using Cepheid Rapid device) will be analysed at ad-hoc exacerbation visits to identify exacerbation pathogenesis.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Respiratory BRU, Nottingham, United Kingdom